CLINICAL TRIAL: NCT05009745
Title: Preimplantation Genetic Testing for Aneuploidy (PGT-A) in in Vitro Fertilisation (IVF) Treatment: Pilot Phase of a Randomised Controlled Trial
Brief Title: Preimplantation Genetic Screening in IVF Treatment
Acronym: PGSINIVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 236067
Record Dates: First submitted 2020-10-28; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Infertility
Keywords: Preimplantation Genetic Testing; IVF; RCT; Pilot Study
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Pilot phase of a prospective, allocation concealed two arm parallel RCT
Masking Description: The participants, care providers, investigators and outcome assessors will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention will be PGT-A strategy involving trophectoderm biopsy and comprehensive chromosome screening (CCS) using Next Generation Sequencing (NGS). All embryos will be frozen after the biopsy procedure and transferred in a subsequent frozen-thawed embryo transfer. Embryo selection for transfer will be based on morphological criteria and the genetic screening result.
  Only euploid embryos or mosaic euploid embryos deemed suitable to be transferred will be replaced into the uterus in a subsequent frozen-thawed embryo transfer cycles.
  Interventions: Procedure: PGT-A Strategy
- Control arm (No Intervention): Women in the control arm will have the fresh embryo transfer procedure on day 5 following egg collection, or a frozen-thawed embryo transfer as first line over a fresh embryo transfer, if clinically indicated. Embryo selection for transfer will be based on morphological criteria.

INTERVENTIONS:
Procedure: PGT-A Strategy — PGT-A strategy involves trophectoderm biopsy, comprehensive chromosome screening (CCS) using Next Generation Screening (NGS), freezing of embryos and replacement in a frozen-thawed embryo transfer cycle.
  Other Names: PGS Strategy
  Arms: Intervention

SUMMARY:
This is the pilot phase of a randomised controlled trial.

The purpose of the pilot study is to assess the ability to recruit, randomise, adherence to the study protocol and plan for a full study.

The purpose of the full study will be to determine if a policy of embryo selection and transfer based on morphological evaluation and preimplantation genetic testing for aneuploidy (PGT-A) is a more clinically effective, safer, cost-effective and acceptable way to provide in vitro fertilisation (IVF) treatment in women of advanced reproductive age compared to the routine practice of embryo selection and transfer based on morphological evaluation alone.

DETAILED DESCRIPTION:
The target population for the trial are women aged 35 - 42 years undergoing IVF±ICSI treatment.

Intervention The experimental strategy will be to perform PGT-A (also referred as preimplantation genetic screening - PGS) involving trophectoderm biopsy on embryos reaching the blastocyst stage on day 5/6/7 following egg collection. All embryos will be frozen after the biopsy procedure.

Comprehensive chromosome screening (CCS) of all chromosomes will be performed using next generation sequencing (NGS). Embryos will be categorised as euploid, mosaic euploid and aneuploid embryos and embryos will be ranked based on the degree of euploidy.

Only euploid embryos or mosaic euploid embryos deemed suitable to be replaced will be transferred in subsequent frozen-thawed embryo transfer cycles.

Comparison Women in the control arm will have the fresh embryo transfer procedure on day 5 following egg collection or a frozen-thawed embryo transfer as first line if clinically indicated in keeping with current routine practice. Embryo selection for transfer will be based on morphological criteria alone.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the study would be women aged 35 - 42 years undergoing IVF ± ICSI for treatment of infertility
* Patients with 3 or more good quality embryos (assessed according to the embryo scoring system of the Association of Clinical Embryologists, UK) on day 3 following egg collection
* Ability to provide informed written consent

Exclusion Criteria:

* Women undergoing preimplantation genetic testing for inherited genetic disorders
* Gamete donation cycles
* Untreated hydrosalpinges
* Untreated uterine pathology (eg: endometrial polyps, submucous fibroids, intramural fibroids > 5 centimetres in maximum diameter, intrauterine adhesions, uterine septa)

Ages: 35 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 18 months
  Pilot phase RCT with an aim to progress to a multi-centre RCT

SECONDARY OUTCOMES:
Clinical pregnancy rate | 21 months
  Clinical pregnancy is defined as presence of an intrauterine gestational sac with a foetal pole and heart beat identified by ultrasound scan.

CONTACTS AND LOCATIONS:
Overall Officials: Sesh K Sunkara, MD, FRCOG, Principal Investigator — King's College London; Ippokratis Sarris, MD, MRCOG, Principal Investigator — King's Fertility, London
Locations (1):
- King's Fertility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
If there was to be an individual participant data (IPD) meta-analysis on this topic or similar collaboration with other researchers in future, we will share IPD with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Beebeejaun Y, Nicolaides KH, Mania A, Sarris I, Sunkara SK. Preimplantation Genetic Testing for Aneuploidy (PGT-A) in In-Vitro Fertilisation (IVF) Treatment: Study Protocol for Pilot Phase of a Randomised Controlled Trial. J Clin Med. 2024 Oct 17;13(20):6192. doi: 10.3390/jcm13206192. PMID 39458142